CLINICAL TRIAL: NCT06469853
Title: A Phase IIa, Open Label, Single Centre Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Orally Dosed MBF-015 in Huntington's Disease Patients
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of MBF-015 in Huntington's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medibiofarma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBF-015CT-02
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBF-015 16 mg oral multiple dose (Experimental): Drug: MBF-015 16 mg oral capsules. Single daily dose. One hard gelatin capsule during 28 days.
  Interventions: Drug: MBF-015 16 mg oral capsules
- MBF-015 32 mg oral multiple dose (Experimental): Drug: MBF-015 16 mg oral capsules. Single daily dose. Two hard gelatin capsules during 28 days.
  Interventions: Drug: MBF-015 16 mg oral capsules

INTERVENTIONS:
Drug: MBF-015 16 mg oral capsules — MBF-015 oral capsules HDAC inhibitor

SUMMARY:
This is a Phase IIa (proof of concept), single center clinical trial to evaluate the safety and efficacy of daily MBF-015 oral treatment during 28 days in Huntington's Disease patients on top of standard of care.

DETAILED DESCRIPTION:
This is a Phase 2a study to evaluate the safety, tolerability and exploratory efficacy of daily oral treatment with either 16 mg or 32 mg MBF-015 during 28 days in Huntington's disease patients with cognitive impairment, in order to provide reliable safety, tolerability, and PK data that will guide drug dose and therapeutic regimen choices in subsequent clinical studies.

The study design is a single-center, open-label group consisting of two cohorts, one dosed with 16 mg MBF-015 daily for 28 days and one dosed with 32 mg MBF-015 daily for 28 days, in approximately 5 subjects per cohort without placebo control. No randomisation is required.

For each subject, the study duration will last a total of approximately 7-9 weeks consisting of a screening period of 1-3 weeks, a treatment period of 4 weeks and a follow-up period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory male or nonpregnant, nonlactating females, age ≥25 to ≤60 years old.
2. Males and females of childbearing potential must agree to use adequate birth control measures during the study. Females of childbearing potential must have a negative serum pregnancy test prior to Visit 2 and either be sexually abstinent or must use a hormonal (oral, implantable, or injectable) or double barrier method of birth control throughout the study, and until 60 days after the last dose of study drug. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or postmenopausal [defined as a minimum of 1 year since the last menstrual period]).
3. Documented CAG triplet repeats ≥39 in the HTT gene. Clinical diagnostic motor features of HD, defined as UHDRS-TMS > 5 with Diagnostic Confidence Score = 4
4. UHDRS Total Functional Capacity (TFC) scores ≥7 and ≤13 with moderate cognitive impairment based on clinical assessment.
5. In the opinion of the Investigator, the patient can tolerate all study procedures and is willing to comply with all other protocol requirements.
6. Able to undergo MRI scans and able to tolerate them (e.g., no metal implants including MRI incompatible IUDs, chorea of a severity that precludes MRI scans or any condition that renders testing intolerable for the patient.
7. Able to tolerate blood draws and lumbar puncture (LP).
8. If participants are using a treatment for HD, they should be on a stable dose for at least 3 months prior to study commencement. Acceptable treatments include Dopamine D2 receptor blockers or reverse agonists, vesicular monoamine transporter 2 blockers or γ-aminobutyric acid (GABA) agonists.
9. Ability to participate fully, in the opinion of the Investigator, in all aspects of this clinical trial. Full comprehension of consent language and written informed consent must be obtained from the participant and documented.

Exclusion Criteria:

1. Clinically significant medical finding on the physical examination other than HD that, in the judgment of the Investigator, will make the patient unsuitable for participation in and/or completion of the study procedures.
2. Clinically significant laboratory abnormality at Screening.
3. Clinically significant abnormality at Screening electrocardiogram (ECG), including but not necessarily limited to a confirmed QT interval corrected for heart rate (QTc) ≥450 msec for males or ≥470 msec for females. Clinically significant cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurologic, malignant, metabolic, psychiatric, or other condition that, in the opinion of the Investigator, precludes the patient's safe participation in the study or would interfere with the study assessments. Mental status, psychiatric medical history, and eligibility for the study must be documented in the screening questionnaire.
4. Pregnant (as determined by a serum pregnancy test) or breast feeding at the Screening Visit, or plans to become pregnant during the course of the study.
5. Deemed to be at significant risk for suicidal behaviour based on any the following criteria:

   1. The opinion of the Investigator
   2. Answers "yes" to Actual Suicide Attempts or Suicidal Behaviors in the Suicidal Behaviors section of the Columbia-Suicide Severity Rating Scale (C-SSRS) with reference to a 2-year period prior to the Screening Visit
   3. Answers "yes" on any items in the Suicidal Ideation section of the C-SSRS with reference to a 6-month period prior to the Screening Visit.
   4. Answers "yes" on any items in the Suicidal Ideation section of the C-SSRS at the Baseline Visit since the last visit (Screening Visit).
6. Positive for Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
7. Known to be positive for human immunodeficiency virus (HIV).
8. Evidence of Clostridioides difficile toxin or treatment for C. difficile infection, or other intestinal bacterial pathogen, within 30 days prior to Screening.Any condition that increases risk of meningitis unless patient is receiving appropriate prophylactic treatment.
9. A medical history of brain or spinal disease that would interfere with lumbar puncture, CSF circulation or safety assessment. History of post-lumbar-puncture headache of moderate or severe intensity and/or blood patch.
10. Contraindication for MRI (claustrophobia, pacemaker, aneurism clips, cardiac mechanical valve).
11. Contraindication for lumbar puncture (anticoagulation, coagulation disease): Must not be taking anticoagulant treatment.
12. Concurrent or previous participation in another clinical trial and received investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to Screening.
13. Any major surgery, in the investigator's opinion, performed within 8 weeks prior to randomization or planned during the study (i.e., any surgical procedure requiring general anesthesia).
14. Unwillingness to withhold protocol-prohibited medications during the trial.
15. Started or changed dose for concomitant medication for the treatment of HD symptoms or psychiatric disorders within 30 days prior to the Screening Visit (concomitant medications that have been administered on a stable regimen for ≥30 days are permitted).
16. History of excessive alcohol or drug abuse that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
17. Positive for opioids (unprescribed), cannabinoids, cocaine, amphetamines, methadone, barbiturates, methamphetamine, or phencyclidine at the Screening Visit.
18. Known or suspected allergy, anaphylaxis, hypersensitivity or intolerance to the study drug excipients.
19. Prior enrolment in the current study and had received study treatment.
20. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 43 days
  Evaluate safety and tolerability of MBF-015 in participants with Huntington's Disease (HD) on top of standard of care over 28 days, with follow-up to day 43.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No